CLINICAL TRIAL: NCT03782766
Title: Mandibular Second Molar Protraction Assisted by and Piezocision
Brief Title: Mandibular Second Molar Protraction Assisted by Piezocision
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jordan University of Science and Technology (Other)
Responsible Party: Principal Investigator, Elham Abu Alhaija, Principal Investigator - Main thesis supervisor, Jordan University of Science and Technology
Allocation: Randomized | Model: Parallel | Purpose: Treatment
Other Study IDs: 416/2016
Record Dates: First submitted 2018-12-15; First posted 2018-12-20 (Actual); Last update posted 2018-12-20 (Actual); Status verified 2018-12

CONDITIONS: Acceleration of Tooth Movement; Piezocision
Keywords: Piezocision; Temporary anchorage device; molar protraction

STUDY DESIGN:
Intervention Model Description: Three models:-
  * Split mouth design where piezocision will be performed on the right of left side of the patient in bilateral first molar extraction space subjects.
  * comparison between 2 groups of subjects; one group where protraction is done with piezocision and the other group where protraction was done with no piezocision.
  * third part where the same side of space receives the 2 interventions. Molar protraction started with no piezocision for 3 months followed by piezocision and protraction for another 3 months,
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- piezosurgery (Experimental): group 1 consisted of 18 molars (13 molars from patients with bilateral first molar extraction space and 5 molars from patients with unilateral first molar extraction space) where piezocesion was performed immediately before molar protraction
  Interventions: Procedure: Piezocision
- No piezocision (No Intervention): group 2 consisted of 21 molars (13 from patients with bilateral first molar extraction space and 8 molars from patients with unilateral first molar extraction space) where molar protraction was performed with no piezocesion
- Late piezocision (Other): group 3 consisted of 21 molars (group 2 subjects where piezocession was carried on after 3 months of molar protraction with no piezocesion.
  Interventions: Procedure: Piezocision

INTERVENTIONS:
Procedure: Piezocision — Piezocesion was performed by making 2 vertical incisions mesial and distal to the extraction space. Piezotome was inserted in the incisions previously made and bone cuts were done with a length up to mucogingival line and depth of 3 mm.
  Arms: Late piezocision; piezosurgery

SUMMARY:
This study was conducted to compare the rate of second molar protraction, level of Interleukin1-β in gingival crevicular fluid, periodontal health (gingival index, plaque index, and periodontal pocket depth) and perception of pain in patients treated by molar protraction with piezocision vs control (no piezocision).

DETAILED DESCRIPTION:
Twenty-six subjects (39 Molars) who presented with at least one extracted mandibular first molar were selected to participate in the study. The subjects were subdivided into one of 3 groups as follows: group 1 consisted of 18 molars (13 molars from patients with bilateral first molar extraction space and 5 molars from patients with unilateral first molar extraction space) where piezocision was performed immediately before molar protraction; group 2 consisted of 21 molars (13 from patients with bilateral first molar extraction space and 8 molars from patients with unilateral first molar extraction space) where molar protraction was performed with no piezocision; group 3 consisted of 21 molars (group 2 subjects where piezocision was carried on after 3 months of molar protraction with no piezocision. After reaching 0.019X0.025" SS arch wire, NiTi coil spring was used for space closure (protraction force was 150g) attached from the lower second molar hook to the head of the mini-screw. Piezocision was performed by making 2 vertical incisions mesial and distal to the extraction space. Piezotome was inserted in the incisions previously made and bone cuts were done with a length up to mucogingival line and depth of 3 mm.

Gingival crevicular fluid (GCF) sample was obtained from the mesiogingival side of the lower second permanent molar with use of Periopaper. GCF sample was repeated 1 day, 1 week and 4 weeks after molar protraction with piezocision or with no piezocision. Pain was assessed using visual analog scale (VAS). Patients were requested to report the level of pain for 7 consecutive days.

ELIGIBILITY:
Inclusion Criteria:

* age range from 20 to 27 years
* at least one extracted mandibular first molar (first molar extracted more than one year ago and residual extraction space more than 5 mm)
* Class 1 malocclusion where molar protraction is indicated
* all permanent teeth are present except for the extracted mandibular first molar/molars.

Exclusion Criteria:-

* Ggingival index score > 2
* Plaque index score > 2
* Probing depth > 4mm
* Previous orthodontic treatment
* Systemic disease and
* Smoker.

Ages: 20 Years to 27 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2015-09-02 (Actual); Primary Completion 2018-10-04 (Actual); Study Completion 2018-10-04 (Actual)

PRIMARY OUTCOMES:
Rate of second molar protraction | up to 3 months
  measured in mm/month from onscreen dental cast
Changes in the level of of Interleukin1-β | Immediately before protraction/piezocision, 1 day, 1 week and 4 weeks after protraction/piezocision
  detected in Gingival crevicular fluid (GCF)

SECONDARY OUTCOMES:
Anchorage loss | Each month up to 3 months
  Distal movement of second premolar in mm per month
Pain Perception: Visual analogue scale (VAS) | Every day up to 7 days
  Assessed using visual analog scale (VAS) where 0 = no pain and 10 = worst pain. The participants filled out questionnaire to assess the pain intensity and interference after second molar protraction with or without piezocision on 1, 2, 3, 4, 5, 6 and 7 days of intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Elham S A Alhaija, Principal Investigator — Prof.- Main thesis supervisor